CLINICAL TRIAL: NCT05034367
Title: Reference Ranges for the Cough Responsiveness to Inhaled Mannitol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kuopio University Hospital (Other)
Collaborators: John Hunter Hospital (Other Government)
Responsible Party: Principal Investigator, Heikki Koskela, Chief physician, Kuopio University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 5801151
Record Dates: First submitted 2021-09-01; First posted 2021-09-05 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Cough
MeSH Terms: conditions — Cough

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Healthy persons (Experimental): The responses of the healthy subjects are utilized to create reference ranges for a normal cough response to mannitol
  Interventions: Diagnostic Test: Mannitol challenge

INTERVENTIONS:
Diagnostic Test: Mannitol challenge — Inhalation challenge with dry powder of mannitol with a maximal cumulative dose of 635 mg

SUMMARY:
Cough is the most common reason why people seek medical attention in developed countries. The main mechanisms for prolonged cough are hypersensitivity of the cough reflex arc, sputum production, and constriction of the airway smooth muscles. Recognition of the mechanism in each cough patient is essential for the efficient management of prolonged cough. At present, there are no feasible tests for everyday clinical work to recognize cough reflex arc hypersensitivity.

Mannitol test was originally developed for asthma diagnostics. We have recently shown that it can also be used to investigate hypersensitive cough reflex arc. The purpose of the present study is to create reference ranges for normal cough responsiveness to inhaled mannitol. Without them, the test cannot be utilized in everyday clinical work. For that purpose we will perform mannitol test in 140 subjects, who are at least 18 years old and without any chronic respiratory symptoms or disorders. The subjects will be recruited in three centers: University of Eastern Finland and: John Hunter Hospital in Australia.The material will be collected 1.9.2021-31.12.2023. We apply funding for both personnel and material expences, to carry out this study.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or older
* capable to understand the purpose of the study
* female/male ratio approximately 50%/50% in both of the following age groups:
* 50% aged 18- 50 yrs, and 50 % aged 51 - 90 years

Exclusion Criteria:

* Current daily smoking
* Ex-smoking with a greater than 10 pack years' daily smoking history or with stopping of daily smoking less than one year ago
* Pregnancy and breastfeeding
* A doctor's diagnosis of any respiratory diseases, including both upper and lower airway diseases, lung parenchymal diseases and the sleep apnoea syndrome
* A doctor's diagnosis of gastro-oesophageal reflux disease or symptoms suggestive of it
* Current use of angiotensin-converting enzyme inhibitors
* Upper respiratory tract infection ('flu') within 4 weeks
* Any current (within 4 weeks) cough 8
* Chronic (over 2 months' duration) cough during the last 12 months
* Wheezing during the last 12 months
* Attacks of shortness of breath or cough at night during the last 12 months
* Symptoms of rhinitis in a prolonged fashion during the last 12 months
* Heartburn or regurgitation once a week or more often during the last 3 months
* Abnormal anatomy of the respiratory organs, which may affect the deposition of the mannitol powder
* Any previous operations to the respiratory organs that can affect the deposition of the mannitol powder
* Unable to provide written informed consent to participate in the study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2022-01-17 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Cough-to-dose ratio | Coughs are recorded during the 60 seconds after each mannitol dose
  calculated as the number of coughs per 100 mg of total cumulative dose of mannitol

CONTACTS AND LOCATIONS:
Locations (2):
- John Hunter Hospital, Newcastle, New South Wales, Australia
- Kuopio University Hospital, Kuopio, Finland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Nurmi HM, Latti AM, Koskela HO. The Cough Response to Inhaled Mannitol in Healthy Subjects. Lung. 2024 Nov 28;203(1):5. doi: 10.1007/s00408-024-00755-6. PMID 39607505